CLINICAL TRIAL: NCT07303491
Title: Translation and Validation of Hindi Version of Oral Health Impact Profile for Chronic Periodontitis (OHIP-CP) a Condition Specific Tool to Assess Oral Health Related Quality of Life in Patients With Chronic Periodontitis
Brief Title: Validation of Hindi Version Oral Health Impact Profile for Periodontitis
Status: Recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: PGIDS/BHRC/25/61
Record Dates: First submitted 2025-11-29; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: OHIP-P-HIN Questionnaire — Hindi Translation of OHIP-CP questionnaire

SUMMARY:
Translation of OHIP-CP questionnaire in Hindi language will be done. Patients recruited will undergo clinical examination and recording of periodontal parameters (Pocket probing Depth and Clinical Attachment Loss) will be recorded to determine stage and grade of periodontitis. Patients will be given OHIP-CP Hindi questionnaire. Content Validity and Construct validity of Hindi translated OHIP-CP questionnaire will be done using appropriate statistical measures. Reliability of the OHIP-CP Hindi questionnaire will be checked for Internal consistency using Cronbach alpha for whole and subscales of OHIP-CP.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* able to understand and complete questionnaires independently
* confirmed diagnosis of periodontitis as defined by the 2017 World Workshop classification.

Exclusion Criteria:

* Patients with systemic diseases such as acquired immunodeficiency syndrome or diabetes mellitus,
* pregnancy
* patients who require prophylactic antibiotic coverage prior to dental treatment,
* patients with bleeding disorders,
* patients had received non-surgical periodontal therapy within the preceding eight weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with periodontitis
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Construct validity | Baseline
  Construct validity of the scale was first evaluated through exploratory factor analysis (EFA) followed by confirmatory factor analysis (CFA)
Reliability Analysis | Baseline
  Internal consistency of the scale will be evaluated using Cronbach's alpha
Discriminant validity | Baseline
  Discriminative validity of the scale will be assessed by comparing mean score differences across varying stages of periodontitis.
Convergent validity | Baseline
  Convergent validity will be evaluated by examining correlations with the global oral health rating.

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS Rohtak, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided